CLINICAL TRIAL: NCT03623009
Title: The Effect of Gender-stigma Consciousness on General Surgery Trainees' Experiences and Skill Performance.
Brief Title: Gender Stigma Consciousness and Surgical Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Sara Myers, UPMC Resident/Fellow, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PRO18040386
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Gender Issues
MeSH Terms: conditions — Sexism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): An article meant to trigger certain psychosocial behaviors is administered to the intervention arm prior to laparoscopic skills assessment.
  Interventions: Behavioral: An article meant to trigger certain psychosocial behaviors
- Control (Sham Comparator): The control arm will receive a neutral article prior to completing the assessment.
  Interventions: Behavioral: a neutral article

INTERVENTIONS:
Behavioral: An article meant to trigger certain psychosocial behaviors — An article meant to trigger certain psychosocial behaviors is administered to the intervention arm prior to laparoscopic skills assessment.
  Arms: Intervention
Behavioral: a neutral article — The control arm will receive a neutral article prior to completing the assessment.
  Arms: Control

SUMMARY:
Previous investigations have focused on challenges that surgeons face once they have entered into practice. We have yet to explore difficulties in the training environment, and whether these have an effect on professional development. In this study, we investigate how certain environmental factors can affect skill acquisition for the resident surgeon. Our trial tests whether psychosocial constructs affect task-performance. This study is a multi-center endeavor with the University of North Carolina-Chapel Hill, the University of Washington, and UPMC. Over an 12 month period, residents will be asked to complete surveys and a laparoscopic skills assessment, which will be administered after residents are randomized to an intervention or control arm. The intervention arm will be asked to read an article that is meant to trigger psychosocial constructs that we hypothesize will affect skill performance. The control arm will receive a neutral article prior to completing the laparoscopic skills assessment.

ELIGIBILITY:
Inclusion Criteria: Categorical General surgery residents who completed undergraduate medical education in the United States

Exclusion Criteria: Residents who have completed graduate medical education training in a subspecialty prior to their general surgery residency.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Score on laparoscopic skills assessment | 12 months
  Score (continuous outcome) based on verified fundamentals of laparoscopic skills assessment grading rubric.

SECONDARY OUTCOMES:
Changes in psychosocial constructs | 12 months
  Changes in Likert scale ratings of psychosocial constructs as assessed by survey with previously published verified sub scales.

CONTACTS AND LOCATIONS:
Overall Officials: Sara P Myers, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Myers SP, Dasari M, Brown JB, Lumpkin ST, Neal MD, Abebe KZ, Chaumont N, Downs-Canner SM, Flanagan MR, Lee KK, Rosengart MR. Effects of Gender Bias and Stereotypes in Surgical Training: A Randomized Clinical Trial. JAMA Surg. 2020 Jul 1;155(7):552-560. doi: 10.1001/jamasurg.2020.1127. PMID 32432669